CLINICAL TRIAL: NCT01143441
Title: Investigating Mechanism of Action of DAC HYP in the Treatment of High-Inflammatory Multiple Sclerosis (MS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100125; 10-N-0125
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2017-08-11

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Daclizumab
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting

ARMS (3):
- Cohort A (Experimental): Long-Term daclizumab cohort
  Interventions: Biological: DAC-HYP
- Cohort B (Experimental): New Treatment Cohort
  Interventions: Biological: DAC-HYP
- Cohort C (No Intervention): MS Controls

INTERVENTIONS:
Biological: DAC-HYP
  Arms: Cohort A; Cohort B

SUMMARY:
Objective:

The primary goal of this study is to investigate the mechanism of action (MOA) of CD25-blocking therapies in high inflammatory multiple sclerosis (HI-MS). The secondary goal of this study is to assess long-term safety and efficacy of CD25-blocking therapies in HI-MS.

Study population:

Two cohorts of patients will be enrolled:

* Long-term daclizumab therapy cohort: Up to 15 daclizumab-treated patients with relapsing-remitting (RR-MS) or secondary-progressive MS (SP-MS) previously classified as HI-MS based on MRI/clinical criteria, who have been treated with IV daclizumab for a minimum of 1 year and responded to this therapy with significant (>70%) decrease in contrast-enhancing lesions (CEL) or stabilization/improvement of disease activity (>60% decrease in MS relapses and stable or improved EDSS disability score).
* New treatment cohort: Up to 15 HI-MS patients (RR- or SP-MS) with inadequate therapeutic response to first-line, FDA-approved immunomodulatory therapies for MS or who cannot, for any reason, be treated with first-line, FDA-approved immunomodulatory therapies for MS.

Design:

This is an open label, Phase I trial of 150 mg of daclizumab high yield process (DAC HYP) administered subcutaneously (SC) every 4 weeks for a total of 3 years.

Outcome measures:

Because the main goal of this study is to investigate the MOA of CD25-blocking therapies in MS, the primary outcomes are mechanistic immunological studies performed on clinical samples (peripheral blood mononuclear cells (PBMC), cerebrospinal fluid (CSF) cells and skin biopsies) derived from DAC HYP-treated patients. The secondary outcome measure is long-term safety and tolerability of subcutaneous DAC HYP in HI-MS patients.

DETAILED DESCRIPTION:
Objective:

The primary goal of this study is to investigate the mechanism of action (MOA) of CD25-blocking therapies in high inflammatory multiple sclerosis (HI-MS). The secondary goal of this study is to assess long-term safety and efficacy of CD25-blocking therapies in HI-MS.

Study population:

We will enroll up to 70 patients. We expect to screen up to 40 HI-MS participants to yield 31 patients that will receive study drug. Two cohorts of patients will be enrolled for the treatment part of the protocol: A. Long-term daclizumab therapy cohort: 16 daclizumab-treated patients with relapsing-remitting (RR-MS) or secondary-progressive MS (SP-MS) previously classified as HI-MS based on MRI/clinical criteria, who have been treated with IV daclizumab for a minimum of 1 year and responded to this therapy with significant (>70%) decrease in contrast-enhancing lesions (CEL) or stabilization/improvement of disease activity (>60% decrease in MS relapses and stable or improved EDSS disability score). B. New treatment cohort: 15 HI-MS patients (RR- or SP-MS) with inadequate therapeutic response to first-line, FDA-approved immunomodulatory therapies for MS or who choose not to, for any reason, be treated with first-line, FDAapproved immunomodulatory therapies for MS. Up to 30 subjects with inflammatory MS will be screened to yield 20 controls for immunization and skin biopsy studies (Cohort C: MS controls).

Design:

This is an open label, Phase I trial of 150 mg of daclizumab high yield process (DAC HYP) administered subcutaneously (SC) every 4 weeks for a total of 3 years.

Outcome measures:

Because the main goal of this study is to investigate the MOA of CD25-blocking therapies in MS, the primary outcomes are mechanistic immunological studies performed on clinical samples (peripheral blood mononuclear cells (PBMC), cerebrospinal fluid (CSF) cells and skin biopsies) derived from DAC HYP-treated patients. The secondary outcome measure is long-term safety and tolerability of subcutaneous DAC HYP in HI-MS patients.

ELIGIBILITY:
* The study population will consist of 2 cohorts of patients with an accrual ceiling of 40 subjects:

A. Long-term daclizumab therapy cohort: Up to 16 patients with HI-MS (both RR-MS and SP-MS) who have been successfully treated with IV daclizumab for a minimum of 1 year.

B. New treatment cohort: Up to 15 patients with HI-MS (both RR-MS and SP-MS) who have not been successfully treated with or have not tolerated standard FDA-approved immunomodulatory therapies, or who, for whatever reason, choose not to be treated with standard FDA approved immunomodulatory therapies.

INCLUSION CRITERIA:

* MS as defined by the modified McDonald criteria (Polman, Reingold et al. 2005)
* HI-MS (RR-MS or SP-MS) before initiation of daclizumab therapy, defined as:

  * greater than or equal to 3 CEL on a single pre-daclizumab MRI or
  * greater than or equal to 1 MS exacerbation per year before initiation of daclizumab therapy or
  * progression of sustained disability by greater than or equal to 1.0 point on the expanded disability status scale (EDSS) in the year preceding daclizumab therapy
  * Age 18-60, inclusive
  * EDSS 0 to 6.0, inclusive
  * Able to provide informed consent
  * Willing to participate in all aspects of trial design and follow-up
  * Females of childbearing potential are willing to commit to the use of a reliable method of birth control (i.e., hormonal contraception including birth control pills, injected hormones or vaginal ring; intrauterine device; barrier methods with spermicide, specifically diaphragms or condoms they have undergone surgical sterilization, such as hysterectomy or tubal ligation) for the duration of the study and continued 4 months after conclusion of the study.

ADDITIONAL INCLUSION CRITERION FOR THE LONG-TERM DACLIZUMAB THERAPY COHORT ONLY:

-IV daclizumab therapy for at least 1 year with a treatment response consisting of:<TAB>

* greater than or equal to 70% reduction of CEL after starting daclizumab; or
* stabilization or improvement of sustained neurological disability on daclizumab.

EXCLUSION CRITERIA (FOR BOTH COHORTS):

* PP-MS or low-inflammatory SP-MS
* Alternative diagnoses that can explain neurological disability and MRI findings (e.g., ischemia/gliosis, CNS lyme disease, SLE, sarcoidosis, etc.)
* History of malignancy, with the following exceptions: excised or treated basal cell carcinoma or fewer than 3 squamous cell carcinomas, grade 1 endometrial carcinomas treated with total hysterectomy and without evidence for recurrence for greater than or equal to 3 years
* Clinically significant medical disorders that, in the judgment of the investigators, could cause CNS tissue damage or limit its repair, expose the patient to undue risk of harm or prevent the patient from completing the study (e.g., immunodeficiency disorders, other autoimmune or immune-mediated disorders or chronic infections). Specific exclusions (based on baseline laboratory evaluation) are:

  * positive HIV or HTLV-1 serology;
  * positive hepatitis B or C serology;
  * pregnant or breastfeeding female;
  * known history of severe allergic or anaphylactic reactions;
  * known hypersensitivity to study drug or its excipients;
  * varicella or herpes zoster virus infection or any severe viral infection within the 6 weeks prior to screening; or
  * exposure to varicella zoster virus within 21 days before screening.
* Abnormal screening/baseline blood tests exceeding any of the limits defined below:

  * serum alanine aminotransferase/serum glutamate pyruvate transaminase (ALT/SGPT), aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT), or gamma-glutamyl-transferase greater than or equal to 2 times the upper limit of normal (ULN);
  * total white blood cell count <3,000/mm(3);
  * hemoglobin greater than or equal to 9.0 g/dL;
  * platelets greater than or equal to 100 x 10(9)/L;
  * lymphocytes greater than or equal to 1.0 x 10(9)/L;
  * neutrophils greater than or equal to 1.5 x 10(9)/L;
  * serum creatinine greater than or equal to the ULN.
* Any of the following treatment history:

  * any type of live virus vaccine in the 4 weeks prior to initiation of therapy, including but not limited to: measles/mumps/rubella vaccine, varicella zoster virus vaccine, oral polio vaccine, and nasal influenza vaccine;
  * infection (viral, fungal, bacterial) requiring hospitalization or intravenous (IV) antibiotics within the 8 weeks prior to initiation of therapy;
  * another investigational drug or approved therapy for investigational use (except daclizumab) within the 6 months prior to initiation of therapy.
* Prior treatment with the any of the following:

  * total lymphoid irradiation;
  * cladribine;
  * T cell or T cell receptor vaccination; or
  * any therapeutic monoclonal antibody, except natalizumab and daclizumab.
* Prior treatment with any of the following medications or procedures within 1 year prior to initiation of therapy:

  * mitoxantrone;
  * cyclophosphamide;
  * fingolimod; or
  * natalizumab.
* Prior treatment with any of the following medications or procedures within 6 months prior to initiation of therapy:

  * cyclosporine;
  * azathioprine;
  * methotrexate;
  * mycophenolate mofetil;
  * intravenous immunoglobulin (IVIg); or
  * plasmapheresis or cytapheresis.
* Treatment with any of the following medications within the 30 days prior to initiation of therapy:

  * IV corticosteroid treatment;
  * oral corticosteroid treatment;
  * glatiramer acetate; or
  * interferon-beta
* For immunizations studies, known history of hypersensitivity or severe allergic reaction to vaccine components (subjects with such history can participate in the trial, but will not be immunized)
* For patients in the extension phase: Patients may be excluded if they did not demonstrate an adequate clinical response in the first phase of the trial while receiving DAC HYP.

Inclusion criteria for MS controls for immunization and skin biopsy studies:

* MS as defined by the modified McDonald criteria
* RR-MS or SP-MS
* Age 18-60, inclusive
* EDSS 0 to 7.0, inclusive
* Able to provide informed consent
* Willing to participate in all aspects of trial design and follow-up

Exclusion criteria for MS controls for immunization and skin biopsy studies:

* Treatment with immunomodulatory therapies that may have a negative impact on development of antigen-specific responses after immunization, including steroids within the last 60 days before the immunization study
* Clinically significant medical disorders that, in the judgment of the investigators, could invalidate the person as appropriate control (e.g., immunodeficiency disorders, other autoimmune or immunemediated disorders or chronic infections). Specific exclusions (based on baseline laboratory evaluation) are:

  * positive HIV or HTLV-1 serology;
  * positive hepatitis B or C serology;
  * pregnant or breastfeeding female;
  * known history of severe allergic or anaphylactic reactions to vaccine components;
* Abnormal screening/baseline blood tests exceeding any of the limits defined below:

  * serum alanine aminotransferase/serum glutamate pyruvate transaminase (ALT/SGPT), aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT), or gamma-glutamyl-transferase (Bullet)2 times the upper limit of normal (ULN);
  * total white blood cell count <3,000/mm3;
  * hemoglobin less than or equal to 9.0 g/dL

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-05-13; Primary Completion 2017-08-11 (Actual); Study Completion 2017-08-11 (Actual)

PRIMARY OUTCOMES:
Expansion of CD56bright NK cells.
Contraction of lymphoid tissue inducer cells (LTi) cells.
Expansion of double negative T cells.

SECONDARY OUTCOMES:
Long-term safety and tolerability of DAC HYP in high-inflammatory multiple sclerosis (HI-MS) patients who were either previously successfully treated with Zenapax (registered trademark) or without any previous exposure to DC25-targeting therapie... | Study Completion
Secondary Outcome Measure: MRI outcomes Inhibition of the number of contrast-enhancing lesions. T2 lesion load and development of new MS lesions. Clinical/functional outcomesChange in EDSS. Change in Scripps NRS. Change in MSFC.Change in S... | Study Completion

CONTACTS AND LOCATIONS:
Overall Officials: Bibiana Bielekova, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bielekova B, Howard T, Packer AN, Richert N, Blevins G, Ohayon J, Waldmann TA, McFarland HF, Martin R. Effect of anti-CD25 antibody daclizumab in the inhibition of inflammation and stabilization of disease progression in multiple sclerosis. Arch Neurol. 2009 Apr;66(4):483-9. doi: 10.1001/archneurol.2009.50. PMID 19364933
- [Background] Hanssen LE, Schrumpf E, Kolbenstvedt AN, Tausjo J, Dolva LO. Recombinant alpha-2 interferon with or without hepatic artery embolization in the treatment of midgut carcinoid tumours. A preliminary report. Acta Oncol. 1989;28(3):439-43. doi: 10.3109/02841868909111219. PMID 2742781
- [Background] Bielekova B, Catalfamo M, Reichert-Scrivner S, Packer A, Cerna M, Waldmann TA, McFarland H, Henkart PA, Martin R. Regulatory CD56(bright) natural killer cells mediate immunomodulatory effects of IL-2Ralpha-targeted therapy (daclizumab) in multiple sclerosis. Proc Natl Acad Sci U S A. 2006 Apr 11;103(15):5941-6. doi: 10.1073/pnas.0601335103. Epub 2006 Apr 3. PMID 16585503